CLINICAL TRIAL: NCT05434780
Title: Comparison of Facilitatory Kinesiology Taping With Combined Inhibitory and Facilitatory Kinesiology Taping Among University Students With Calf Tightness
Brief Title: Kinesiology Taping on Calf Tightness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSAHS 2022/001
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Calf Muscle Pulled
Keywords: Kinesiology Taping, Calf Tightness, Ankle ROM and Balance

STUDY DESIGN:
Intervention Model Description: 20 consented subjects will be randomly divided into 2 equal groups using goldfish bowl method.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After getting the consent, baseline measurements will be taken by the assessor. An assessor performing the tests will be blind to the assigned intervention to avoid expectation bias.After taking baseline measurements, all twenty participants will be given a fictitious number and according to these numbers subjects will be allocated to two different groups using Goldfish Bowl randomization method. Ten participants will be allocated to group A in which facilitatory taping will be applied on the calf muscles and the other ten will be allocated in group B in which inhibitory K Tape will be applied to calf muscles and facilitatory K taping will be applied on Tibialis anterior muscle. KT will be applied by a physiotherapist who will be blind to the purpose of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Intervention 1 or group A) (Active Comparator): Facilitatory kinesiology taping on calf muscles
  Interventions: Other: Kinesiology taping
- (Intervention 2 or group B) (Experimental): Inhibitory kinesiology taping on calf Muscles combined with Facilitatory kinesiology taping on Tibialis Anterior
  Interventions: Other: Kinesiology taping

INTERVENTIONS:
Other: Kinesiology taping — Kinesiology tape is an elastic tape applied to skin with specific amount of tension as per requirement. The underlying mechanism investigated by several studies is the space enhancement and skin uplifting that increases the blood flow in the targeted area and promotes healing.

SUMMARY:
This study aims to determine the effect of combined facilitatory Kinesiology and inhibitory Kinesiology taping on balance and ROM in university students with calf tightness. This study will also compare Inhibitory kinesiology taping on calf muscles with combined Inhibitory and Facilitatory kinesiology taping on tight Calf and weak Tibialis anterior respectively This randomized clinical trial will include 20 university students with calf tightness according to inclusion and exclusion criteria. Subjects will be assessed by using silfverskiold test for calf tightness and star excursion test for dynamic balance. Baseline measurements will be documented and the subjects will be randomly assigned to two interventions by Goldfish Bowl randomization method: Facilitatory kinesiology taping on calf muscles (Intervention 1 or group A) and Inhibitory kinesiology taping on calf Muscles combined with Facilitatory kinesiology taping on Tibialis Anterior (Intervention 2 or group B). Immediate effects of taping on balance will be assessed after 20 minutes. After that follow up will be maintained and participants will be assessed again after 72 hours. At the end, these measurements will be documented and compared with baseline readings. And changes will be noted down. The data will be entered and analyzed using SPSS 25.

DETAILED DESCRIPTION:
Leg pain is considered one of the most common issues worldwide. It can be due to variety of factors like medial tibial stress syndrome, nerve compression, overuse, musculoskeletal disorders and arterial or venous disorders. According to the literature, muscle tightness is one of the most common factors responsible for leg pain.The area most prone to muscle tightness in lower limb is lower leg region specifically calf muscles. Calf tightness is a common problem in healthy population especially students who have to sit for prolong durations. Studies have reported venous insufficiency causing calf pain in female university students who wear high heels on habitual basis.

Prevalence of calf pain in patients with Ankle foot pathologies is 96.5%. For example, patients with talipes equinus, Achilles tendinopathies, metatarsalgia and mid foot arthritis present with restricted ankle ROM and pain in calf region. Certain systemic diseases can also cause calf tightness like, peripheral vascular disease, Deep Venous Thrombosis, muscle strain or tendon injuries. It can vary from mild to intense. It can be symptomatic (bruising, swelling or sudden pain) or asymptomatic. Furthermore, it has been shown to be a significant factor in postural and balance dysfunction accompanied by proprioception problems. Disturbed balance and proprioception can be attributed to decreased dorsiflexion range of motion that is basically a consequence of over activity of calf muscles.

Different strategies have been used to treat calf tightness that include RICE (Rest, Ice Compression Elevation) protocol, stretching, ankle mobilization, Proprioceptive Neuromuscular Facilitation, electrotherapy, soft tissue mobilization, Taping and other manual therapy techniques. Taping has remained really an effective treatment to release calf tightness. Literature has shown remarkable effects of Kinesiology Tape application in variety of musculoskeletal conditions like, plantar fasciitis, ankle sprain, medial tibial stress syndrome, general knee pain and low back pain.

Kinesiology tape is an elastic tape applied to skin with specific amount of tension as per requirement. The underlying mechanism investigated by several studies is the space enhancement and skin uplifting that increases the blood flow in the targeted area and promotes healing. According to the recent studies, kinesiology Taping significantly support weak muscles, decrease pain by lifting fascia, helps to reposition subluxated joint as well as enhance muscle function by increasing strength and proprioception.

As existing literature provide evidence, KT improves healing by fastening tissue repair and increasing vascularity. It can be attributed to increased amount of type III collagen fibers as documented in a recent study. A recent study conducted in 2021 on comparison between the conservative treatment and combined effects of KT with conservative treatment showed significant improvements in healing.KT has also remained an efficacious treatment for hallux valgus patients as it decreases the hallux angle and pain.

In addition to its effects in musculoskeletal conditions, KT has played significant role in lymphatic drainage and swelling or edema reduction. Tape is applied in a fan shaped pattern and the strips are called fan shaped strips or edema strips. According to a previous study, KT combined with manual lymphatic drainage significantly decreased the post-operative lymphedema in breast surgery patients than using manual lymphatic techniques only. Studies have been conducted that support the idea that KT plays a significant role in injury protection and prevention in sports. Moreover, its role in stroke is undeniably important causing improved integration of the three systems that maintain stability i.e. motor, sensory and CNS integration.

Different application methods of K Taping have been used in management of Soft Tissue Injuries. K Tape effectiveness mainly relies on its direction of application and its shapes as well. Shapes used can be I, Y, X, web or donut shaped. Applied direction effect has been used to achieve the desired function of KT that can be facilitation or inhibition of muscles. Taping from origin to insertion can be used to facilitate the weak muscles while taping from insertion to origin can be used to inhibit the over active or spastic muscles.

Conditions like scapula-thoracic dysfunction cause hyperactivity of the upper fibers of the trapezius which can be treated by using inhibitory kinesiology taping. It has been also very effective in treating the hyperactivity of vastas lateralis to treat patellofemoral pain syndrome and lateral patellar tracking. This inhibitory effect can be attributed to shortening effect of tape that decreases the tonic discharge and causes relaxation. In a recent study conducted on chronic stroke patients, two types of taping PNF-KT and A-KT were applied and significant increase in ankle dorsiflexion ROM and balance was observed but PNF-KT more significantly improved ankle DF-ROM and static balance than A-KT.The use of inhibitory kinesiology taping alone can also be used in chronic stroke patients to decrease the over activity of spastic muscles. In another study conducted on the comparison of effects of direction of application of kinesiology tape on sensation and postural control, improvement in sensation and sway speed was observed with facilitatory and inhibitory taping respectively. Furthermore facilitation taping improved two-point discrimination and increased the sensitivity of combined cortical sensation

Literature supports the use of either facilitatory or inhibitory taping on a certain muscle but no evidence to the best of researcher knowledge exists in literature supporting the simultaneous use of Inhibitory taping on tight muscles and Facilitatory Taping on Weak muscles. Furthermore the combined effect of Inhibitory and Facilitatory Taping on Balance and ankle ROM in Adults with Calf Tightness is still unclear. So, this study aims to evaluate the combined effect of simultaneous application of inhibitory taping on tight calf and facilitatory taping on tibialis anterior and how it improves balance and ROM.

Purpose of this study is to devise more efficient and time saving treatment strategy for clinicians and healthcare professionals. This study will help to improve Balance and Range of Motion in adults with calf tightness by comparing the effects of two Taping Strategies. This study will reduce the cost and time of patients by giving them better management option using Kinesiology Taping leading to fast recovery as well as reducing the risk of injuries and further complications.

ELIGIBILITY:
Inclusion Criteria:

* Both Male & Female
* Age between 18 to 28 years old university students with Calf Tightness.

Exclusion Criteria:

* Students with plantar fascitis, history of fractures, bone spurs, any arthritis, any history of pain, trauma, or injury of the knee joint, triceps surae muscles or ankle joint 6 months prior to the study.
* Skin disease or self-reported hypersensitivity to tape application, including scar tissue in the acute phase.
* Any red flag (rheumatoid arthritis, metabolic diseases, psychological problem, fibromyalgia, Spinal fracture, previous spinal trauma, tumor etc) or subjects with chronic illness (musculoskeletal, systemic, psychological or any comorbidity i.e. diabetes, hypertension, hematological issues, etc

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Ankle Range of Motion | 72 Hours of Treatment
  Ankle Range of Motion in individuals with Calf Tightness will be measured by Silfverskiold test

SECONDARY OUTCOMES:
Dynamic Balance | 72 Hours of Treatment.
  Dynamic Balance in Individuals with calf Tightness will be assessed by Star excursion test

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Fiza, DPT, Principal Investigator — Shalamar Institute of Health Sciences; Rommana Zubair, DPT, Principal Investigator — Shalamar Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park D, Bae Y. Proprioceptive Neuromuscular Facilitation Kinesio Taping Improves Range of Motion of Ankle Dorsiflexion and Balance Ability in Chronic Stroke Patients. Healthcare (Basel). 2021 Oct 22;9(11):1426. doi: 10.3390/healthcare9111426. PMID 34828473
- [Background] Ataullah MG, Kapoor G, Alghadir AH, Khan M. Effects of kinesio taping on hip abductor muscle strength and electromyography activity in athletes with chronic ankle instability: A randomized controlled trial. J Rehabil Med. 2021 Jun 4;53(6):jrm00204. doi: 10.2340/16501977-2845. PMID 34013356
- [Background] Tomruk MS, Tomruk M, Alkan E, Gelecek N. Is Ankle Kinesio Taping Effective to Immediately Change Balance, Range of Motion, and Muscle Strength in Healthy Individuals? A Randomized, Sham-Controlled Trial. Korean J Fam Med. 2022 Mar;43(2):109-116. doi: 10.4082/kjfm.21.0015. Epub 2022 Mar 17. PMID 35320896
- [Background] Arshad Z, Aslam A, Razzaq MA, Bhatia M. Gastrocnemius Release in the Management of Chronic Plantar Fasciitis: A Systematic Review. Foot Ankle Int. 2022 Apr;43(4):568-575. doi: 10.1177/10711007211052290. Epub 2021 Nov 12. PMID 34766860
- [Background] Li Y, Liu X, Luo X, Guo C. Effect of Tai Chi combined with Kinesio taping on posture control of football players with FAI: protocol for a randomized controlled trial. Trials. 2022 Feb 19;23(1):162. doi: 10.1186/s13063-022-06083-5. PMID 35183232
- [Background] Landorf KB, Kaminski MR, Munteanu SE, Zammit GV, Menz HB. Clinical measures of foot posture and ankle joint dorsiflexion do not differ in adults with and without plantar heel pain. Sci Rep. 2021 Mar 19;11(1):6451. doi: 10.1038/s41598-021-85520-y. PMID 33742026